CLINICAL TRIAL: NCT04370938
Title: Exploring Provider Burnout During the COVID-19 Pandemic
Brief Title: Provider Burnout During COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled and the study was never initiated.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sara Myers, General Surgery Residents, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY20040051
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Perceived Organizational Support, Anxiety, Burnout
MeSH Terms: conditions — Anxiety Disorders; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: A longitudinal survey-based research study investigating the domains of perceived organizational support, anxiety, and burnout will take place. Healthcare providers with patient-care contact will be asked to fill out these surveys once every 30 days over a period of 6 months. After the first survey is complete, 20% of participants will be randomized to watch a 1-hour long video discussing coping strategies for stress related to the COVID-19 pandemic.
Who Masked: Outcomes Assessor
Masking Description: Individuals responsible for analyzing survey data (including that which was administered after the intervention), will be masked with regard to whether the participant received the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coping strategies video (Experimental): Individuals will be asked to watch a 1 hour long video that discusses strategies helpful in coping with stress during the COVID-19 pandemic.
  Interventions: Behavioral: Coping strategies video
- Control (No Intervention): No additional requests will be made of individuals in the control arm.

INTERVENTIONS:
Behavioral: Coping strategies video — No additional description
  Arms: Coping strategies video

SUMMARY:
Since the novel coronavirus, SARS-CoV-2, was first reported in the Hubei province of China in December 2019, the US has become an epicenter for the pandemic, accounting for more than 220,000 cases and 4,800 deaths (CDC). The rapid spread of the associated disease, COVID-19, has overwhelmed healthcare systems in spite of unprecedented measures to reduce contagion. The resulting uncertainty with regard to the duration and magnitude of the pandemic and limited availability of resources and treatment have been detrimental to the mental health of frontline healthcare providers (NIH). Preserving the psychological wellbeing of these individuals is paramount to mitigating the effect of COVID-19 and delivering optimal patient care.

Of particularly grave concern is how professional and personal distress caused by the COVID-19 pandemic will affect provider burnout (Lai et al. JAMA Network Open 2020). Professional burnout, characterized by emotional exhaustion, career de-prioritization, and loss of self-efficacy, represents a significant threat to the US healthcare system (Shanafelt et al. Ann Surg 2010; Han et al. Annals of Internal Medicine 2019). While burnout has been described as a reaction to chronic work-related stress (Melamed et al. Psychol. Bull. 2006), individual factors such as anxiety increase susceptibility to burnout (Sun et al. J Occup Health 2012). Although data suggests that occupational stress might amplify risk of anxiety (DiGiacomo and Adamson J Allied Health 2001), we have yet to understand how intensified anxiety among frontline providers during global health crises contributes to burnout. Similarly, it is unknown whether factors such as perceived organizational support (POS), a key driver of job satisfaction and performance (Muse and Stamper, J Managerial Issues 2007), modify anxiety and burnout under these circumstances. We hypothesize that diminished POS in response to the COVID-19 pandemic is associated with burnout and that this relationship is mediated by an increase in providers' anxiety. Delineating this relationship is a critical first step in developing interventions that ease the mental health burden of this pandemic and future crises for healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* All UPMC healthcare providers with patient-care responsibilities (respiratory therapists, physical therapists, nursing staff, residents, attendings, midlevel providers, and clinical faculty) will be contacted via email and asked if they would be willing to participate in this study (participant recruitment email).

Exclusion Criteria:

* All individuals <18 yo and those providers without direct patient-care responsibilities will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-10-29 (Estimated); Study Completion 2020-10-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility of undertaking task | 6 months
  As healthcare providers have limited time, it is unclear if this request to watch a 1 hour video on coping strategies will be a feasible intervention. We will assess how many individuals endorse actually watching this video.

CONTACTS AND LOCATIONS:
Overall Officials: Sara P Myers, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided